CLINICAL TRIAL: NCT07147114
Title: A Multicenter, Randomized, Double-Blind, Exploratory Clinical Trial to Evaluate the Efficacy and Safety in Concomitant Administration of Macitentan and Dapagliflozin in Patients With Heart Failure With Mildly Reduced and Preserved Ejection Fraction (HFmrEF and HFpEF) and Combined Pre- and Post-capillary Pulmonary Hypertension (CpcPH)
Brief Title: Clinical Trial to Evaluate the Efficacy and Safety in Concomitant Administration of Macitentan and Dapagliflozin in Patients With Heart Failure With Mildly Reduced and Preserved Ejection Fraction (HFmrEF and HFpEF) and Combined Pre- and Post-capillary Pulmonary Hypertension (CpcPH)
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Gachon University Gil Medical Center (Other)
Responsible Party: Principal Investigator, Wook-Jin Chung, Principal Investigator, Gachon University Gil Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MD-CpcPH
Record Dates: First submitted 2025-08-21; First posted 2025-08-28 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Combined Pre- and Post-capillary Pulmonary Hypertension; CpcPH; HFmrEF; HFpEF; Group 2 Pulmonary Hypertension
MeSH Terms: interventions — Combined Modality Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combination therapy group (Experimental): Maciten Tab. 10mg
  Interventions: Drug: Combination therapy
- Monotherapy group (Placebo Comparator): Dapozin Tab. 10mg or 5mg
  Interventions: Drug: Monotherapy

INTERVENTIONS:
Drug: Combination therapy — Macitentan 10mg, Dapagliflozin 10mg or 5mg po tablet q.d. in 24 weeks
  Other Names: Maciten Tab. 10mg
  Arms: Combination therapy group
Drug: Monotherapy — Macitentan placebo, Dapagliflozin 10mg or 5mg po tablet q.d. in 24 weeks
  Other Names: Dapozin Tab. 10mg or 5mg
  Arms: Monotherapy group

SUMMARY:
This clinical trial will evaluate whether combination therapy with Dapagliflozin + Macitentan improves outcomes compared to Dapagliflozin + placebo in patients with combined pre- and post-capillary pulmonary hypertension (CpcPH).

The study will measure changes in pulmonary vascular resistance, NT-proBNP, 6-minute walk distance, and quality of life (KCCQ scores) over 24 weeks.

Participants will be randomly assigned to one of two groups, take study medication for 24 weeks, and undergo regular clinical, laboratory, and safety assessments.

ELIGIBILITY:
Inclusion Criteria:

<Screening Visit (Visit 1)>

1. A male or female adults aged 19 years or older in South Korea
2. LVEF greater than 40% on echocardiogram performed within 12 weeks prior to screening
3. Presence of heart failure with mildly reduced ejection fraction (HFmrEF) or preserved ejection fraction (HFpEF) accompanied by combined pre- and post-capillary pulmonary hypertension (CpcPH)
4. Meeting all of the following criteria on RHC performed within 48 weeks prior to screening:

   1. mPAP > 20 mmHg
   2. PVR > 2 Wood units (WU)
   3. PAWP > 15 mmHg
5. World Health Organization Functional Class (WHO-FC) II or III at the time of screening
6. If taking any of the following medications at the time of screening, the participant must have been on a stable dose for at least 3 months:

   1. Renin-angiotensin system inhibitors
   2. Beta-blockers
   3. Mineralocorticoid receptor antagonists (aldosterone antagonists)
   4. Sodium-glucose cotransporter-2 (SGLT2) inhibitors
   5. Ivabradine

<Baseline Visit (Visit 2)>

1. World Health Organization Functional Class (WHO-FC) II or III at the time of baseline visit

Exclusion Criteria:

<Screening Visit (Visit 1)>

1. Known hypersensitivity to the active ingredients (Macitentan, Dapagliflozin) or any excipients of the investigational medicinal product
2. Pregnant or breastfeeding women, or those who do not agree to use at least two appropriate contraceptive methods* (self or partner) during the clinical trial period and for 30 days after the last administration of the investigational medicinal product (for male participants, those who do not agree to refrain from sperm donation)

   *: a. Surgical sterilization (e.g., vasectomy) or intrauterine device (IUD; copper IUD or hormone-releasing intrauterine system), b. Non-oral hormonal contraceptive or spermicide in combination with a barrier method, c. Cervical cap or diaphragm used in combination with a male condom.
3. Participants with type 1 diabetes mellitus or secondary diabetes mellitus
4. Participants with metabolic acidosis, such as diabetic ketoacidosis
5. Participants diagnosed with pulmonary hypertension other than WHO Group 2 pulmonary hypertension (i.e., WHO Group 1, 3, 4, or 5)

   1. Group 1: Pulmonary arterial hypertension
   2. Group 3: Pulmonary hypertension associated with lung diseases and/or hypoxia
   3. Group 4: Chronic thrombo-embolic pulmonary hypertension
   4. Group 5: Pulmonary hypertension with unclear and/or multifactorial mechanisms
6. Participants who meet the following criteria on RHC performed within 48 weeks prior to screening:

   a. PAWP ≤ 15 mmHg
7. History of taking any of the following medications within 4 weeks prior to screening:

   1. Calcium channel blockers
   2. Endothelin receptor antagonists
   3. Phosphodiesterase type 5 inhibitors (PDE5i)
   4. Riociguat, Vericiguat
   5. Prostacyclin (PC) analogs or prostacyclin receptor agonists
   6. Activin signaling inhibitors
8. History of any of the following medical conditions, surgeries, or procedures:

   1. Myocardial infarction, coronary artery bypass grafting, or percutaneous coronary intervention (PCI) within 3 months prior to screening
   2. Uncontrolled tachycardia (>110 bpm) due to atrial fibrillation or atrial flutter
   3. History of heart transplantation or implantation of a ventricular assist device, or planned to undergo such procedures
9. eGFR ≤ 30 mL/min/1.73 m² or AST or ALT ≥ 2.5 × ULN
10. Urinary tract infection, genital infection (including fungal infections), or voiding disorder within 24 weeks prior to screening
11. Hemoglobin < 9 g/dL at the time of screening
12. Participants with genetic disorders such as galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption
13. Known hypersensitivity to soybean oil or history of soybean oil allergy
14. Known hypersensitivity to soy or peanuts
15. Participation in another clinical trial involving administration/application of an investigational medicinal product or medical device within 3 months prior to screening

<Baseline Visit (Visit 2)>

1. Participants who, upon re-confirmation of inclusion/exclusion criteria at the baseline visit, have any disqualifying condition
2. Any other condition that, in the opinion of the investigator, makes the participant unsuitable for participation in this clinical trial

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-10-31 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Hierarchical outcome component(Change in PVR, Change in NT-proBNP, Change in 6MWD, Change in KCCQ-CSS) | Baseline, 24 week
  The hierarchical composite variable includes the rate of change in Pulmonary Vascular Resistance (PVR), NT-proBNP, change in 6-minute walk distance, and change in KCCQ-CSS score. All possible pairwise comparisons between combination therapy group and monotherapy group subjects (e.g., 2 subjects in combination group and 3 in monotherapy group yield 6 pairs) are classified as Win, Loss, or Tie based on the following definitions. If the subject in the pair meeting the criteria belongs to the combination group, it is evaluated as a Win; if in the monotherapy group, a Loss.

SECONDARY OUTCOMES:
Change in Pulmonary Vascular Resistance (PVR) from Baseline to Week 24 | Baseline, 24 week
  PVR (Wood Units, WU) is measured by Right Heart Catheterization (RHC).
Change in Mean Pulmonary Arterial Pressure (mPAP) from Baseline to Week 24 | Baseline, 24 week
  mPAP (mmHg) is measured by RHC.
Change in Pulmonary Arterial Wedge Pressure (PAWP) from Baseline to Week 24 | Baseline, 24 week
  PAWP (mmHg) is measured by RHC.
Change in 6-Minute Walk Distance from Baseline to Week 24 | Baseline, 24 week
  Distance (meters) measured by 6-minute walk test.
Change in Oxygen Saturation (SpO2) Difference Before and After 6-Minute Walk Test from Baseline to Week 24 | Baseline, 24 week
  Oxygen saturation (%) difference before and after the 6-minute walk test.
Change in N-terminal pro-brain natriuretic peptide (NT-proBNP) from Baseline to Week 24 | Baseline, 24 week
  NT-proBNP (pg/mL) measured by clinical laboratory tests.
Change in Tricuspid Regurgitation Velocity (TRV) from Baseline to Week 24 | Baseline, 24 week
  TRV (m/s) measured by echocardiography.
Change in Tricuspid Annular Plane Systolic Excursion (TAPSE) from Baseline to Week 24 | Baseline, 24 week
  TAPSE (mm) measured by echocardiography.
Use of Intravenous Diuretics During Treatment Period (Visit 2 to Visit 4) | Baseline, 24 week
  The number of intravenous diuretic administrations collected via concomitant medication records.
Rate of Hospitalization Due to Heart Failure During Treatment Period (Visit 2 to Visit 4) | Baseline, 24 week
  Number of hospitalizations for heart failure compared between groups during treatment period.
Number of Days Hospitalized for Heart Failure During Treatment Period (Visit 2 to Visit 4) | Baseline, 24 week
  Total days of hospitalization for heart failure compared between groups during treatment.
Number of Deaths (Cardiovascular and All-Cause) During Treatment Period (Visit 2 to Visit 4) | Baseline, 24 week
  Cardiovascular and all-cause mortality events compared between groups.
Change in Mean Right Atrial Pressure (mRAP) from Baseline to Week 24 | Baseline, 24 week
  mRAP (mmHg) measured by RHC.
Change in Cardiac Index (CI) from Baseline to Week 24 | Baseline, 24 week
  Cardiac Index (L/min/m²) measured by RHC.
Change in Mixed Venous Oxygen Saturation (SvO2) from Baseline to Week 24 | Baseline, 24 week
  SvO2 (%) measured by RHC.
Change in Left Atrial Volume Index (LAVI) from Baseline to Week 24 | Baseline, 24 week
  LAVI (mL/m²) measured by echocardiography and body measurements.
Change in Tricuspid Valve Systolic Tissue Velocity (TV S' velocity) from Baseline to Week 24 | Baseline, 24 week
  TV S' velocity (cm/s) measured by echocardiography.
Change in Right Atrial Area (RA area) from Baseline to Week 24 | Baseline, 24 week
  RA area (cm²) measured by echocardiography.
Change in Presence of Pericardial Effusion from Baseline to Week 24 | Baseline, 24 week
  Presence or absence of pericardial effusion evaluated by echocardiography.
Change in Kansas City Cardiomyopathy Questionnaire Overall Summary Score (KCCQ-OSS) from Baseline to Week 24 | Baseline, 24 week
  KCCQ-OSS measured by questionnaire.

CONTACTS AND LOCATIONS:
Locations (15):
- South Korea (15):
  - Pusan National University Hospital, Busan
  - Chungbuk National University Hospital, Chungju
  - Keimyung University Dongsan Hospital, Daegu
  - Chungnam National University Hospital, Daejeon
  - Chonnam National University Hospital, Gwangju
  - Incheon Sejong Hospital, Incheon
  - Gachon University Gil Hospital, Incheon
  - Seoul National University Hospital, Seoul
  - Yonsei University Health System, Severance Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea, Seoul St.Mary, Seoul
  - Koera University Guro Hospital, Seoul
  - Yonsei University, Wonju Severance Christian Hospital, Wŏnju
  - Pusan National University Yangsan Hospital, Yangsan

IPD SHARING:
Plan to Share IPD: No